CLINICAL TRIAL: NCT05129436
Title: Blood Donations From Healthy Volunteers for the Study of the Adaptive Immune Response to Seasonal Influenza Vaccination (AIGI)
Brief Title: Adaptive Immune Response to Seasonal Influenza Vaccination (AIGI)
Acronym: (AIGI)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: AIGI
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Seasonal Influenza Vaccination
Keywords: vaccine; vaccination; seasonal influenza; influenza; immune response; immunokinetics
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Establishment of method: healthy volunteers who are asked to donate peripheral blood for the establishment of the method
- Influenza vaccination: Subjects receiving the influenza vaccine Vaxigrip Tetra 2020/2021 by Sanofi Pasteur Europe.
  Interventions: Drug: Vaxigrip Tetra 2020/2021

INTERVENTIONS:
Drug: Vaxigrip Tetra 2020/2021 — vaccine against seasonal influenza
  Groups: Influenza vaccination

SUMMARY:
AIGI (Adaptive Immune Response to Seasonal Influenza Vaccination) is a prospective clinical study aiming at studying the kinetics of vaccine-specific antibody production after seasonal influenza vaccination in health care workers.

DETAILED DESCRIPTION:
AIGI (Adaptive Immune Response to Seasonal Influenza Vaccination) is a prospective clinical study aiming at elucidating the kinetics of vaccine-specific antibody production after seasonal Influenza vaccination in health care workers at the Greifswald University hospital. Participants were recruited before their intended vaccination.

Participants received the influenza vaccine Vaxigrip Tetra 2020/2021 by Sanofi Pasteur Europe.

Within the study, volunteers donate peripheral blood by venipuncture on the day of vaccination as well as 7 and 14 days after vaccination. EDTA plasma and peripheral mononuclear cells (PBMCs) are prepared and stored at -20 °C.

Volunteers are also asked to complete a standardized questionnaire on each day of blood sampling. Questionnaires collect data about physical characteristics, seasonal influenza vaccinations, current infections, medication, immune relevant diseases and side effects of the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Planned participation in seasonal influenza vaccination
* Completion of the 18th year of life
* verbal and written consent given

Exclusion Criteria:

* current infectious diseases
* underweight (BMI<18,5)
* blood coagulation disorders, anemia or similar diseases
* known congenital or acquired immunodeficiencies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Employees at the University Medicine Greifswald, Germany, who plan to be vaccinated against seasonal influenza
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mean current anti-influenza antibody production and cumulative antibody titer on the day of the vaccination | 1 day
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts.
  For this purpose PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted on the day of the vaccination.
mean current anti-influenza antibody production 7 days after the vaccination | 7 days after the vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 7 days after the vaccination.
mean current anti-influenza antibody production 14 days after the vaccination | 14 days after the vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 14 days after the vaccination.

SECONDARY OUTCOMES:
plasma antibody levels against seasonal influenza | 3 weeks
  anti-influenza antibodies are quantified using ELISA
immune cell phenotyping (B cells, T cells) | 3 weeks
  flow cytometry-based analyses

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M. Bröker, Prof. Dr., Study Chair — University Medicine Greifswald, Dept. of Immunology
Locations (1):
- University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Undecided